CLINICAL TRIAL: NCT07358585
Title: A Phase Ib/II Study to Evaluate the Efficacy, Safety and Tolerance of HLX43 (an Anti-PD-L1 Antibody Conjugated) Combined With HLX07 (a Recombinant Anti-EGFR Humanized Monoclonal Antibody) or Serplulimab in Patients With Advanced or Metastatic Colorectal Cancer
Brief Title: A Phase Ib/II Study to Evaluate HLX43 Combined With HLX07 or Serplulimab in Patients With Advanced or Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-mCRC202
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms | interventions — HLX07

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HLX43 dose 1 (Experimental): HLX43 dose 1 + HLX07 1000mg, Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 1 + HLX07
- HLX43 dose 2 (Experimental): HLX43 dose 2 + HLX07 1000mg, Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 2 + HLX07
- HLX43 dose 3 (Experimental): HLX43 dose 3 + Serplulimab 300mg, Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 3 + Serplulimab
- HLX43 dose 4 (Experimental): HLX43 dose 4 + Serplulimab 300mg, Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 4 + Serplulimab

INTERVENTIONS:
Drug: HLX43 dose 1 + HLX07 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  HLX07 is a recombinant anti-EGFR humanized monoclonal antibody
  Arms: HLX43 dose 1
Drug: HLX43 dose 2 + HLX07 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  HLX07 is a recombinant anti-EGFR humanized monoclonal antibody
  Arms: HLX43 dose 2
Drug: HLX43 dose 3 + Serplulimab — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Serplulimab is an anti-PD-1 humanized monoclonal antibody
  Arms: HLX43 dose 3
Drug: HLX43 dose 4 + Serplulimab — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Serplulimab is an anti-PD-1 humanized monoclonal antibody
  Arms: HLX43 dose 4

SUMMARY:
This study is a phase Ib/II study to evaluate the efficacy, safety and tolerance of HLX43 combined with HLX07 or Serplulimab in patients with advanced or metastatic colorectal cancer failed or intolerance to standard first-line therapy

DETAILED DESCRIPTION:
This study is a phase Ib/II study to evaluate the efficacy, safety and tolerance of HLX43 (an Anti-PD-L1 antibody conjugated) combined with HLX07 (a recombinant anti-EGFR humanized monoclonal antibody) or Serplulimab in patients with advanced or metastatic colorectal cancer failed or intolerance to standard first-line therapy In this study, eligible subjects will be randomized at 1:1 ratio in 2 different groups in 2 parts (part HLX43 + HLX07 and part HLX43 + Serplulimab) . The patients will be administered with HLX43 at different doses combined with HLX07 or Serplulimab via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced or metastatic colorectal adenocarcinoma; and locally tested and confirmed as a RAS/BRAF wild-type tumor (only for Part 1 );
2. Previously failed first-line systemic anti-tumor therapy for advanced or metastatic colorectal adenocarcinoma based on a 5-FU regimen, with radiologically documented disease progression.

   Note: For patients who have previously received radical concurrent chemoradiotherapy, neoadjuvant/adjuvant chemotherapy, or chemoradiotherapy, if disease progression occurred during treatment or within ≤6 months after treatment cessation, it should be considered as first-line treatment failure; if progression occurred beyond 6 months, it should not be considered as first-line treatment failure.
3. Patients known to have dMMR/MSI-H must have failed treatment containing a PD-1 immune checkpoint inhibitor, with radiologically documented disease progression (only for Part 1);
4. There must be an interval of at least 4 weeks or 5 half-lives of the drug (whichever is longer) from the first dose of the investigational drug to prior major surgery, medical device treatment, local radiotherapy (except palliative radiotherapy for bone metastases), cytotoxic chemotherapy, macromolecular targeted drug therapy, immunotherapy, or biologic therapy; an interval of at least 2 weeks from prior small molecule targeted drug therapy; an interval of at least 1 week from prior traditional Chinese medicine therapy with anti-tumor indications or minor surgery; and all prior anti-tumor treatment-related adverse events (AEs) must have recovered to CTCAE v5.0 Grade ≤1 (except peripheral neuropathy and alopecia).
5. Adequate organ function.

Exclusion Criteria:

1. Prior exposure to any drug targeting topoisomerase I, including chemotherapy or antibody-drug conjugates (ADCs); prior treatment with anti-EGFR antibody therapy (only for Part 1); prior treatment with PD-1/PD-L1 inhibitors or any immunotherapy targeting immune checkpoints (only for Part 2).
2. Candidates suitable for locoregional treatment with curative intent (e.g., surgery or radiotherapy).
3. History of a second malignant neoplasm within 2 years prior to randomization, except for early-stage malignancies treated with curative intent (e.g., carcinoma in situ or Stage I tumors), such as non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer, ductal carcinoma in situ of the breast, or papillary thyroid cancer.
4. Known or suspected history of keratitis, ulcerative keratitis, or severe dry eye disease.
5. History of adverse events leading to permanent discontinuation of prior immunotherapy; or history of ≥ Grade 2 immune-mediated pneumonitis or immune-mediated myocarditis.
6. Use of strong inhibitors or inducers of CYP2D6 or CYP3A within 2 weeks prior to randomization.
7. Active HBV or HCV infection or co-infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-07-28 (Estimated); Study Completion 2028-08-23 (Estimated)

PRIMARY OUTCOMES:
ORR | From enrollment to 12 weeks after last patient in
  Objective response rate (ORR) (assessed by BICR according to the RECIST v1.1 criteria)
PFS | rom date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by BICR according to the RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China